CLINICAL TRIAL: NCT06306326
Title: Application of Three-dimensional Facial Scanning Images in Evaluating the Therapeutic Efficacy of Autologous Fat Grafting in the Treatment of Craniofacial Deformities
Brief Title: 3D Facial Scanning for Evaluating Autologous Fat Grafting in Craniofacial Deformities
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pkussfatgrafting
Record Dates: First submitted 2024-02-27; First posted 2024-03-12 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-02

CONDITIONS: Adipocytes; Autografts; Imaging, Three-Dimensional / Methods
Keywords: Autologous Fat Grafting; 3dMD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D Facial Scanning for Evaluating Autologous Fat Grafting in Craniofacial Deformities (Experimental): By performing autologous fat grafting surgery on 100 patients with craniofacial deformities that meet the research criteria, 3dMD technology will be used for facial three-dimensional scanning preoperatively, immediately postoperatively, and at six months postoperatively to obtain facial volume data. Then, through precise data analysis, we will calculate the fat absorption rate and study the effects of individual factors on treatment outcomes through correlation regression analysis.
  Interventions: Diagnostic Test: 3dMD technology

INTERVENTIONS:
Diagnostic Test: 3dMD technology — By taking photos using 3dMD, we obtained preoperative, immediate postoperative, and long-term postoperative three-dimensional data of patients. The software automatically fused the data to obtain the volume difference of facial volume at different time points, and then divided it to obtain the objective data of facial volume improvement rate. To improve the reliability of the measurements, two researchers measured independently and took the average value.

SUMMARY:
Treatment of craniofacial deformities is a significant topic in oral and maxillofacial surgery, and autologous fat grafting has become one of the main methods for treating facial concave deformities. However, the instability of its treatment effect has always been a bottleneck in this field, mainly due to the uncertain absorption rate of transplanted fat. This project aims to use advanced the 3dMD face system (3dMD) (3dMD Inc, Atlanta, Ga) technology to precisely measure the facial volume changes before and after autologous fat grafting to address this issue. By performing autologous fat grafting surgery on 100 patients with craniofacial deformities that meet the research criteria, 3dMD technology will be used for facial three-dimensional scanning preoperatively, immediately postoperatively, and at six months postoperatively to obtain facial volume data. Then, through precise data analysis, we will calculate the fat absorption rate and study the effects of individual factors on treatment outcomes through correlation regression analysis.

DETAILED DESCRIPTION:
Craniofacial deformities are common facial abnormalities that can significantly affect patients' appearance and oral function, leading to profound impacts on their psychological and quality of life. Autologous fat grafting has been used since the early 20th century for facial filling, offering advantages such as using the patient's own tissues, minimal risk of rejection, and providing a natural appearance. Therefore, it has become a popular method in plastic surgery and widely used to treat various types of facial deformities. However, the technique also presents clinical challenges, as the transplanted fat cells need sufficient blood supply in the new location to survive and maintain their volume. During the process, a portion of the transplanted fat tissue without blood supply will be absorbed. Generally, the absorption rate of transplanted fat tissue varies from 30% to 70% depending on factors such as location, surgical technique, time, and individual differences, leading to unstable outcomes. Factors affecting the survival rate of fat particles after transplantation include infection, poor blood supply in the recipient area, age, physique, nutrition, mental state, and the duration of the deformity. Shallow depressions have a lower absorption rate, while deeper ones have a higher absorption rate. Postoperative immobilization of the transplanted fat area is necessary to rebuild blood circulation. However, there is no literature reporting the exact impact of these factors on the absorption rate of fat grafts. Therefore, it is suggested that autologous fat grafting should be performed using the "small amount multiple times" method for timely correction.

In addition to being influenced by surgical techniques and individual differences, a more significant issue is the lack of accuracy in assessing the effectiveness of this technique. Previous evaluation methods include subjective assessment and objective evaluation methods such as cephalometric measurements. However, these methods have various degrees of inaccuracy in evaluating soft tissue volume changes. The emergence of the 3dMD face system (3dMD) (3dMD Inc, Atlanta, Ga) technology is expected to solve this problem. 3dMD technology, full name 3D facial scanning imaging technology, uses binocular vision principles to rapidly capture three-dimensional data of the face, providing high-precision facial morphology information. It is accurate, fast, and radiation-free, and literature suggests it is the preferred method for evaluating the results of facial soft tissue volume recovery surgery. The application of 3dMD technology can help achieve precise measurements of facial volume before and after fat grafting, providing a powerful tool for studying fat absorption rates.

This study is an observational study that will use 3dMD technology to accurately measure changes in facial volume before and after autologous fat grafting by scanning the patient's face in three dimensions. This will provide accurate fat absorption or retention rates and study the impact of individual factors on treatment outcomes through regression analysis. This will help better understand the effectiveness of autologous fat grafting technology and provide a scientific basis for the treatment of craniofacial deformities.

ELIGIBILITY:
Inclusion Criteria:

* Facial soft tissue volume deficiency deformity caused by congenital/acquired factors, meeting the indications for autologous fat grafting surgery.
* Good physical health, without severe systemic diseases or infectious diseases.
* Not pregnant and without plans for pregnancy.
* Signed informed consent form.

Exclusion Criteria:

* Contraindications to general anesthesia.
* Patient refusal to participate in this study.
* Significant contour changes in non-filled facial areas during follow-up period leading to inability to register data.

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Fat Retention Rate | 4 weeks postoperative and 1 year postoperative.
  Using 3dMD technology, facial profiles were captured preoperatively and postoperatively. The postoperative profiles were matched with the preoperative ones and processed using Boolean operations to obtain the volume difference, which represents the volume of grafted fat. The fat retention rate was calculated by dividing the volume of grafted fat obtained at 1 year postoperatively by the volume obtained at 1 month postoperatively.

SECONDARY OUTCOMES:
Patient Satisfaction | 4 weeks postoperative and 1 year postoperative.
  Patient satisfaction with the improvement in facial appearance was assessed using a Visual Analog Scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Xi Gong, Dr, Study Director — Peking University School and Hospital of Stomatology

IPD SHARING:
Plan to Share IPD: No